CLINICAL TRIAL: NCT07061808
Title: The Reliability and Validity of the Turkish Version of the Lipedema Screening Questionnaire
Brief Title: The Reliability and Validity of the Turkish Version of the LSQ
Acronym: LSQ
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ilke Keser, Proffesor, Gazi University
Other Study IDs: Canan Lipedema Screening Q.
Record Dates: First submitted 2025-06-14; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Lipedema; Women
Keywords: lipedema; validity; reliability; Turkish adaptation
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women diagnosed with lipoedema: women diagnosed with lipoedema
  Interventions: Diagnostic Test: Lipedema Screening Questionnaire

INTERVENTIONS:
Diagnostic Test: Lipedema Screening Questionnaire — The Lipoedema screening questionnaire (LSQ) is a practical tool that can be applied quickly and easily and is used to identify patients with lipoedema during history taking and physical examination.

SUMMARY:
Abstract Background/ Aim: The aim of this study was to investigate the reliability and validity of the Turkish version of the Lipedema Screening Questionnaire (T-LSQ). Method: The study involved 59 female volunteers diagnosed with lipedema by a cardiovascular surgeon. Key demographics such as age, onset age, lipedema types and stages, clinical features, and BMI were recorded. The Turkish adaptation of the LSQ was performed in accordance with the protocol of Beaton. Confirmatory factor analysis was performed for structural validity. For concurrent validity, T- LSQ, the Lower Extremity Functional Scale (LEFS), the Lymphedema Life Impact Scale (LLIS), and the Lymphoedema Functioning, Disability and Health Quastionnaire for Lower Extremity Lymphedema (Lymph-ICF-LL) were applied and the correlation between the scale responses was analyzed. Test-retest and internal consistency reliability were performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* had no communication cognitive and mental problem
* participant in Turkish

Exclusion Criteria:

* Patients with diagnoses of renal and heart failure
* individuals with history of lower extremity surgery
* individuals with severe arterial venous disease involving the lower extremity
* individuals with active cancer disease or metastasis
* individuals with severe acute infective disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Lipedema is a disease that usually affects women. Lipedema affects approximately 11% of the female population and its aetiology has not yet been elucidate.
Study Population: Information provided about the study and informed consent was obtained from voluntary participants. Participants who came to University hospital physiotherapy department for treatment or control purposes with the diagnoses of lipoedema, lipolymphoedema were included in the study.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
The Validity and Reliability of Turkish version of the Lipedema Screening Questionnaire | at 10-day intervals.
  The Validity and Reliability of Turkish version of the Lipedema Screening Questionnaire: For validity, T-LSQ, Lower Extremity Functional Scale (LEFS), Lymphedema Life Impact Scale (LLIS) and Lymphedema Function, Disability and Health Questionnaire for Lower Extremity Lymphedema (Lymph-ICF-LL) were applied and correlation analysis between scale responses will be done. The LSQ questionnaire, whose reliability we measured, was applied at the beginning of the study and again after 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- aDepartment of Physiotherapy and Rehabilitation, Health Science Faculty, Gazi University, Ankara, Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't feel the need to.

REFERENCES:
- [Result] Devoogdt N, Van Kampen M, Geraerts I, Coremans T, Christiaens MR. Lymphoedema Functioning, Disability and Health questionnaire (Lymph-ICF): reliability and validity. Phys Ther. 2011 Jun;91(6):944-57. doi: 10.2522/ptj.20100087. Epub 2011 Apr 14. PMID 21493748
- [Result] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Result] Herbst KL, Kahn LA, Iker E, Ehrlich C, Wright T, McHutchison L, Schwartz J, Sleigh M, Donahue PM, Lisson KH, Faris T, Miller J, Lontok E, Schwartz MS, Dean SM, Bartholomew JR, Armour P, Correa-Perez M, Pennings N, Wallace EL, Larson E. Standard of care for lipedema in the United States. Phlebology. 2021 Dec;36(10):779-796. doi: 10.1177/02683555211015887. Epub 2021 May 28. PMID 34049453
- [Result] Mishra, Manit. (2016). Confirmatory Factor Analysis (CFA) as an Analytical Technique to Assess Measurement Error in Survey Research: A Review. Paradigm. 20. 97-112. 10.1177/0971890716672933.
- [Result] Zinbarg, R.E., Revelle, W., Yovel, I. et al. Cronbach's α, Revelle's β, and Mcdonald's ω H : their relations with each other and two alternative conceptualizations of reliability. Psychometrika 70, 123-133 (2005). https://doi.org/10.1007/s11336-003-0974-7
- [Result] Feise RJ, Michael Menke J. Functional rating index: a new valid and reliable instrument to measure the magnitude of clinical change in spinal conditions. Spine (Phila Pa 1976). 2001 Jan 1;26(1):78-86; discussion 87. doi: 10.1097/00007632-200101010-00015. PMID 11148650
- [Result] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Result] Citaker S, Kafa N, Hazar Kanik Z, Ugurlu M, Kafa B, Tuna Z. Translation, cross-cultural adaptation and validation of the Turkish version of the Lower Extremity Functional Scale on patients with knee injuries. Arch Orthop Trauma Surg. 2016 Mar;136(3):389-95. doi: 10.1007/s00402-015-2384-6. Epub 2016 Jan 4. PMID 26728274
- [Result] Degirmenci B, Tuzun S, Of NS, Oral A, Sindel D. Reliability and validity of Turkish version of Lymphedema Life Impact Scale. Turk J Phys Med Rehabil. 2019 May 3;65(2):147-153. doi: 10.5606/tftrd.2019.3041. eCollection 2019 Jun. PMID 31453555
- [Result] Kostanoglu A, Hosbay Z, Tarakci E. Lymphoedema functioning, disability and health questionnaire Turkish version: translation, cross-cultural adaptation and validation. J Phys Ther Sci. 2016 Jun;28(6):1728-32. doi: 10.1589/jpts.28.1728. Epub 2016 Jun 28. PMID 27390404
- [Result] Begum, M. R. (2019). Validity and Reliability of Visual Analogue Scale (Vas) for Pain Measurement.
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Weiss J, Daniel T. VALIDATION OF THE LYMPHEDEMA LIFE IMPACT SCALE (LLIS): A CONDITION-SPECIFIC MEASUREMENT TOOL FOR PERSONS WITH LYMPHEDEMA. Lymphology. 2015 Sep;48(3):128-38. PMID 26939160
- [Result] Devoogdt N, De Groef A, Hendrickx A, Damstra R, Christiaansen A, Geraerts I, Vervloesem N, Vergote I, Van Kampen M. Lymphoedema Functioning, Disability and Health Questionnaire for Lower Limb Lymphoedema (Lymph-ICF-LL): reliability and validity. Phys Ther. 2014 May;94(5):705-21. doi: 10.2522/ptj.20130285. Epub 2014 Jan 10. PMID 24415775
- [Result] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Result] Kerola T, Hiltunen M, Kettunen R, Hartikainen S, Sulkava R, Vuolteenaho O, Nieminen T. Mini-Mental State Examination score and B-type natriuretic peptide as predictors of cardiovascular and total mortality in an elderly general population. Ann Med. 2011 Dec;43(8):650-9. doi: 10.3109/07853890.2010.526137. Epub 2010 Oct 21. PMID 20961273
- [Result] Meier-Vollrath I, Schmeller W. [Lipoedema--current status, new perspectives]. J Dtsch Dermatol Ges. 2004 Mar;2(3):181-6. doi: 10.1046/j.1439-0353.2004.04051.x. German. PMID 16281634
- [Result] Nuttall FQ. Body Mass Index: Obesity, BMI, and Health: A Critical Review. Nutr Today. 2015 May;50(3):117-128. doi: 10.1097/NT.0000000000000092. Epub 2015 Apr 7. PMID 27340299
- [Result] Herbst KL. Rare adipose disorders (RADs) masquerading as obesity. Acta Pharmacol Sin. 2012 Feb;33(2):155-72. doi: 10.1038/aps.2011.153. PMID 22301856
- [Result] WOLD LE, HINES EA Jr, ALLEN EV. Lipedema of the legs; a syndrome characterized by fat legs and edema. Ann Intern Med. 1951 May;34(5):1243-50. doi: 10.7326/0003-4819-34-5-1243. No abstract available. PMID 14830102
- [Result] Czerwinska M, Teodorczyk J, Hansdorfer-Korzon R. A Scoping Review of Available Tools in Measurement of the Effectiveness of Conservative Treatment in Lipoedema. Int J Environ Res Public Health. 2022 Jun 10;19(12):7124. doi: 10.3390/ijerph19127124. PMID 35742373
- [Result] Kruppa P, Georgiou I, Biermann N, Prantl L, Klein-Weigel P, Ghods M. Lipedema-Pathogenesis, Diagnosis, and Treatment Options. Dtsch Arztebl Int. 2020 Jun 1;117(22-23):396-403. doi: 10.3238/arztebl.2020.0396. PMID 32762835
- [Result] Szolnoky G, Nagy N, Kovacs RK, Dosa-Racz E, Szabo A, Barsony K, Balogh M, Kemeny L. Complex decongestive physiotherapy decreases capillary fragility in lipedema. Lymphology. 2008 Dec;41(4):161-6. PMID 19306662
- [Result] Buck DW 2nd, Herbst KL. Lipedema: A Relatively Common Disease with Extremely Common Misconceptions. Plast Reconstr Surg Glob Open. 2016 Sep 28;4(9):e1043. doi: 10.1097/GOX.0000000000001043. eCollection 2016 Sep. PMID 27757353
- [Result] Reich-Schupke S, Schmeller W, Brauer WJ, Cornely ME, Faerber G, Ludwig M, Lulay G, Miller A, Rapprich S, Richter DF, Schacht V, Schrader K, Stucker M, Ure C. S1 guidelines: Lipedema. J Dtsch Dermatol Ges. 2017 Jul;15(7):758-767. doi: 10.1111/ddg.13036. PMID 28677175
- [Result] Katzer K, Hill JL, McIver KB, Foster MT. Lipedema and the Potential Role of Estrogen in Excessive Adipose Tissue Accumulation. Int J Mol Sci. 2021 Oct 29;22(21):11720. doi: 10.3390/ijms222111720. PMID 34769153
- [Result] Amato ACM, Amato FCM, Benitti DA, Amato LGL. Development of a questionnaire and screening model for lipedema. J Vasc Bras. 2020 Dec 11;19:e20200114. doi: 10.1590/1677-5449.200114. PMID 34211528
- [Result] Shavit E, Wollina U, Alavi A. Lipoedema is not lymphoedema: A review of current literature. Int Wound J. 2018 Dec;15(6):921-928. doi: 10.1111/iwj.12949. Epub 2018 Jun 29. PMID 29956468
- [Result] Child AH, Gordon KD, Sharpe P, Brice G, Ostergaard P, Jeffery S, Mortimer PS. Lipedema: an inherited condition. Am J Med Genet A. 2010 Apr;152A(4):970-6. doi: 10.1002/ajmg.a.33313. PMID 20358611
- See also: Related Info — https://wounds-uk.com/wp-content/uploads/2023/02/450f55130cff87901188206fd115ccf3.pdf
- See also: Related Info — https://library.lipedema.org/bibliography/2NJUI9JP
- See also: Related Info — https://www.researchgate.net/publication/237524921_Estimating_Generalizability_to_a_Latent_Variable_Common_to_All_of_a_Scale's_Indicators_A_Comparison_of_Estimators_for_h
- See also: Related Info — https://search.trdizin.gov.tr/tr/yayin/detay/19471/standardize-mini-mental-test-in-turk-toplumunda-hafif-demans-tanisinda-gecerlik-ve-guvenilirligi